CLINICAL TRIAL: NCT00728936
Title: A Phase 1, Multi-center, Placebo-controlled, Dose-escalation Study of the Safety of IMO-2125 in Hepatitis C-infected Patients Unresponsive to Standard Treatment With Pegylated Interferon and Ribavirin
Brief Title: Placebo-controlled, Dose-escalation Study of the Safety of IMO-2125 (Immunomodulatory Oligonucleotide) in Hepatitis C-infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idera Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMO-2125-001
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2017-11

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; unresponsive to pegylated interferon and ribavirin therapy; hepatitis C virus
MeSH Terms: conditions — Hepatitis C | interventions — tilsotolimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- IMO-2125 0.04 mg/kg q week (Experimental): IMO-2125 given weekly at 0.04 mg/kg
  Interventions: Drug: IMO-2125
- IMO-2125 0.08 mg/kg q week (Experimental): IMO-2125 given weekly at 0.08 mg/kg
  Interventions: Drug: IMO-2125
- IMO-2125 0.16 mg/kg q week (Experimental): IMO-2125 given weekly at 0.16 mg/kg
  Interventions: Drug: IMO-2125
- IMO-2125 0.32 mg/kg q week (Experimental): IMO-2125 given weekly at 0.32 mg/kg
  Interventions: Drug: IMO-2125
- IMO-2125 0.48 mg/kg q week (Experimental): IMO-2125 given weekly at 0.48 mg/kg
  Interventions: Drug: IMO-2125
- Placebo (Placebo Comparator): Weekly saline placebo
  Interventions: Drug: Saline placebo
- IMO-2125 0.16 mg/kg twice a week (Experimental): IMO-2125 given twice a week at 0.16 mg/kg
  Interventions: Drug: IMO-2125

INTERVENTIONS:
Drug: IMO-2125 — IMO-2125 is a synthetic DNA-based agonist of Toll-like receptor 9 (TLR9), TLR9 is expressed in humans in plasmacytoid dendritic cells and B cells of the immune system
  Arms: IMO-2125 0.04 mg/kg q week; IMO-2125 0.08 mg/kg q week; IMO-2125 0.16 mg/kg q week; IMO-2125 0.16 mg/kg twice a week; IMO-2125 0.32 mg/kg q week; IMO-2125 0.48 mg/kg q week
Drug: Saline placebo — saline placebo given subcutaneously
  Arms: Placebo

SUMMARY:
First-in-humans, phase 1, dose-escalation study with 4 dose levels of single-agent IMO-2125.

DETAILED DESCRIPTION:
First-in-humans, phase 1, dose-escalation study with 4 dose levels of single-agent IMO-2125. Patients will proceed through a screening period, treatment period, and follow-up period of approximately 4 months' duration. There will be 4 dose cohorts including active drug and placebo dosing.

ELIGIBILITY:
Inclusion Criteria:

* HCV-positive
* Nonresponder to standard-dose pegylated interferon-α-2a or -α-2b in combination with standard-dose ribavirin

Exclusion Criteria:

* Human immunodeficiency virus (HIV)or hepatitis B surface antigen (HbsAg)
* Inadequate bone marrow, liver, and renal function
* Treatment with any IFN (interferon)-based or other experimental or antiviral therapies within 30 days
* Other significant medical diseases
* Known alcohol or drug abuse within the past 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Bexon, MD, Study Director — Idera Pharmaceuticals
Locations (7):
- United States (6):
  - University of Colorado Hospital, Aurora, Colorado
  - Gastoenterstinal Specialist of Georgia, PA, Marietta, Georgia
  - Henry Ford Med Ctr- Columbus, Novi, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - The Liver Institute, Dallas, Texas
  - Alamo Medical Research, San Antonio, Texas
- Fundacion de Investigacion de Diego, Santurce, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled patients with chronic infection with hepatitis C virus (HCV) who were "null responders" to prior treatment with pegylated-interferon-alfa (peg-IFN-α) plus ribavirin. The study included patients with any HCV genotype.
Pre-assignment Details: All enrolled subjects who qualified after the pre-screening period were assigned to a treatment group and treated.
Period: Overall Study
Arm/Group | Placebo | IMO-2125 0.04 mg/kg q Week | IMO-2125 0.08 mg/kg q Week | IMO-2125 0.16 mg/kg q Week | IMO-2125 0.32 mg/kg q Week | IMO-2125 0.48 mg/kg q Week | IMO-2125 0.16 mg/kg Twice a Week
Started | 10 | 8 | 9 | 8 | 8 | 8 | 7
Completed | 10 | 8 | 9 | 8 | 8 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | IMO-2125 0.04 mg/kg q Week | IMO-2125 0.08 mg/kg q Week | IMO-2125 0.16 mg/kg q Week | IMO-2125 0.32 mg/kg q Week | IMO-2125 0.48 mg/kg q Week | IMO-2125 0.16 mg/kg Twice a Week | Total
Number analyzed (Participants) | 10 | 8 | 9 | 8 | 8 | 8 | 7 | 58
Age, Continuous [Median (Full Range); unit: years] | 50 [43 to 57] | 55 [45 to 59] | 51 [30 to 61] | 55.5 [50 to 65] | 49 [42 to 55] | 52.5 [35 to 58] | 56 [19 to 63] | 54 [30 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 2 | 1 | 1 | 0 | 1 | 15
  Male | 4 | 4 | 7 | 7 | 7 | 8 | 6 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 4 | 2 | 2 | 0 | 11
  White | 8 | 7 | 9 | 4 | 6 | 6 | 6 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HCV Genotype [Count of Participants; unit: Participants]
  1a | 7 | 4 | 6 | 6 | 4 | 7 | 4 | 38
  1b | 3 | 3 | 3 | 2 | 4 | 1 | 3 | 19
  4a or 4c or 4d | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Safety.
Description: Count and percentage of subjects with treatment emergent adverse events
Time Frame: From screening through study completion, 86 to 115 days in total
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | IMO-2125 0.04 mg/kg q Week | IMO-2125 0.08 mg/kg q Week | IMO-2125 0.16 mg/kg q Week | IMO-2125 0.32 mg/kg q Week | IMO-2125 0.48 mg/kg q Week | IMO-2125 0.16 mg/kg Twice a Week
Number analyzed (Participants) | 10 | 8 | 9 | 8 | 8 | 8 | 7
Participants
  At least 1 TEAE | 6 | 8 | 9 | 8 | 8 | 8 | 7
  Study drug-related TEAE | 5 | 7 | 9 | 8 | 8 | 8 | 7
  TEAE leading to study drug discontinuation | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Related TEAE causing study drug discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious Adverse Events | 0 | 0 | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: From screening through study completion, 86 to 115 days in total
Description: Any untoward medical occurrence in a clinical investigation patient administered a pharmaceutical product; it does not necessarily have to have a causal relationship with this treatment. An Adverse Event can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporarily associated with the use of a medicinal product, whether or not considered to be related to the medicinal product.
Arm/Group | Placebo | IMO-2125 0.04 mg/kg q Week | IMO-2125 0.08 mg/kg q Week | IMO-2125 0.16 mg/kg q Week | IMO-2125 0.32 mg/kg q Week | IMO-2125 0.48 mg/kg q Week | IMO-2125 0.16 mg/kg Twice a Week
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/9 | 0/8 | 0/8 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/9 | 0/8 | 0/8 | 1/8 | 0/7
Other Adverse Events (participants affected / at risk) | 6/10 | 8/8 | 9/9 | 8/8 | 8/8 | 8/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | IMO-2125 0.04 mg/kg q Week (N=8) | IMO-2125 0.08 mg/kg q Week (N=9) | IMO-2125 0.16 mg/kg q Week (N=8) | IMO-2125 0.32 mg/kg q Week (N=8) | IMO-2125 0.48 mg/kg q Week (N=8) | IMO-2125 0.16 mg/kg Twice a Week (N=7)
Erosive esophaghitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | IMO-2125 0.04 mg/kg q Week (N=8) | IMO-2125 0.08 mg/kg q Week (N=9) | IMO-2125 0.16 mg/kg q Week (N=8) | IMO-2125 0.32 mg/kg q Week (N=8) | IMO-2125 0.48 mg/kg q Week (N=8) | IMO-2125 0.16 mg/kg Twice a Week (N=7)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastric mucosal lesion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hiatis hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoasethsia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 2 | 2 | 3
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Chills (General disorders) | 0 | 0 | 2 | 2 | 3 | 2 | 1
Fatigue (General disorders) | 1 | 3 | 1 | 2 | 2 | 1 | 2
Influenza-like illness (General disorders) | 2 | 5 | 5 | 4 | 4 | 7 | 5
Injection site dermatitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 1 | 5 | 9 | 8 | 8 | 8 | 7
Injection site hematoma (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 3
Injection site hemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Injection site induration (General disorders) | 1 | 5 | 6 | 4 | 7 | 7 | 6
Injection site edema (General disorders) | 1 | 1 | 3 | 0 | 1 | 1 | 0
Injection site pain (General disorders) | 1 | 1 | 2 | 4 | 3 | 5 | 6
Injection site paraesthesia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritis (General disorders) | 1 | 4 | 1 | 2 | 4 | 2 | 2
Injection site rash (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site warmth (General disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 4
Edema peripheral (General disorders) | 1 | 1 | 0 | 1 | 4 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 1 | 4 | 1 | 0
Injection site cellulitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 1 | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 2 | 2 | 0 | 1
Headache (Nervous system disorders) | 2 | 2 | 0 | 4 | 5 | 2 | 3
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes